CLINICAL TRIAL: NCT00110903
Title: Open-Label Study to Assess the Safety of Etanercept Liquid Administered Once Weekly in Subjects With Active Rheumatoid Arthritis (RA)
Brief Title: Treatment for Subjects With Active Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20020378
Record Dates: First submitted 2005-05-16; First posted 2005-05-17 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; RA; etanercept; Immunex; Amgen
MeSH Terms: conditions — Arthritis, Rheumatoid

INTERVENTIONS:
Drug: Etanercept Liquid

SUMMARY:
The purpose of this study is to assess the safety of etanercept liquid administered once weekly to subjects with RA.

ELIGIBILITY:
Inclusion Criteria: - Fulfill the 1987 American Rheumatism Association (ARA) criteria for RA - Active RA at the time of enrollment, receipt of concomitant methotrexate at a dose of up to 25 mg a week is permitted - Screening lab results must demonstrate:

* AST and ALT less than or equal to 2 times the upper limit of normal hemoglobin greater than or equal to 8.5 g/dL;
* Platelet count greater than or equal to 125,000/cm3;
* White blood cell count (WBC) greater than or equal to 3500 cells/cm3;
* Serum creatinine less than or equal to 2 mg/dL - Before any study specific procedure is performed, the subject must provide informed consent for participation in the study Exclusion Criteria: - Previous receipt of etanercept - Receipt of antibody to (tumor necrosis factor) TNF alpha or other TNF inhibitors within 90 days of Day 1 - Currently enrolled in other investigational device or drug trials, or participation in investigational trial within the past 30 days - Receipt of intra-articular corticosteroids within 14 days prior to Day 1 - Receipt of any disease-modifying anti-rheumatic drugs (DMARDs) within 28 days of Day 1 - Receipt of cyclophosphamide within 6 months of Day 1 - Concomitant corticosteroids greater than 10 mg/day of prednisone (or equivalent) during 14 days prior to Day 1 - Dose of nonsteroidal anti-inflammatory drug (NSAID) must be stable for 14 days prior to Day 1 and must not exceed the recommended dose in the product information sheet - Subject is not using adequate contraception - Subject is pregnant or breast-feeding - Subject has significant concurrent medical disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Proportion of subjects having positive immunoassay response to etanercept liquid during the treatment period.

SECONDARY OUTCOMES:
Incidence of adverse events, infectious episodes, serious adverse events, serious infectious episodes
Measurements from safety laboratory assessments.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Dore RK, Mathews S, Schechtman J, Surbeck W, Mandel D, Patel A, Zhou L, Peloso P. The immunogenicity, safety, and efficacy of etanercept liquid administered once weekly in patients with rheumatoid arthritis. Clin Exp Rheumatol. 2007 Jan-Feb;25(1):40-6. PMID 17417989
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com